CLINICAL TRIAL: NCT02293057
Title: Gender-Responsive Drug Use Treatment for Juvenile Justice Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA035231-01A1 (NIH)
Record Dates: First submitted 2014-10-31; First posted 2014-11-18 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Drug Use
Keywords: Adolescent; Juvenile Justice; Drug Use; Marijuana; Gender Responsive; Girls; HIV; Sexual Risk
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VOICES Group (Active Comparator): VOICES: A program of self-discovery and empowerment includes four modules: Self (A), Connecting with others (B), Healthy living (C), and the Journey Ahead (D). All sessions are 60 minutes long and include required and optional activities.
  Interventions: Behavioral: VOICES Group
- Girl Health Group (Attention Control) (Placebo Comparator): The Girl Health group comparison condition includes adolescent groups matched for time and attention to VOICES groups. Intervention take a psychoeducational/didactic approach and content focuses on a range of health behaviors, including substance use, exercise, nutrition and sleep.
  Interventions: Behavioral: Girl Health Group

INTERVENTIONS:
Behavioral: VOICES Group — VOICES: A program of self-discovery and empowerment includes four modules: Self (A), Connecting with others (B), Healthy living (C), and the Journey Ahead (D). All sessions are 60 minutes long and include required and optional activities.
  Arms: VOICES Group
Behavioral: Girl Health Group — The Girl Health group comparison condition includes adolescent groups matched for time and attention to VOICES groups. Intervention take a psychoeducational/didactic approach and content focuses on a range of health behaviors, including substance use, exercise, nutrition and sleep.
  Arms: Girl Health Group (Attention Control)

SUMMARY:
Girls in the juvenile justice system have unique developmental pathways to drug use and co-occurring risk (e.g., HIV/STI) behaviors that have typically not been considered or tested in order to identify evidence-based gender-specific substance use treatment approaches for this population. This study will advance scientific knowledge and clinical practice in the drug treatment and public health fields by testing the efficacy of a pre-existing, widely disseminated gender-responsive substance use treatment (VOICES) on drug use and HIV/STI risk behavior outcomes for a broad range of substance using girls and young women (ages 12-24) who are at-risk for or already involved with the justice system.

DETAILED DESCRIPTION:
Compared to both non-offending females and male offending counterparts, offending girls are at significantly greater risk for the development of substance use disorders, psychiatric symptoms and negative health outcomes, such as HIV/AIDS or other sexually transmitted infections (STIs). Research suggests that girls may have different developmental pathways to drug use, initial legal involvement and co-occurring negative health outcomes that support the importance of testing gender-specific treatments for juvenile justice girls. Although there is recent increased emphasis on gender-specific programming in juvenile justice, empirically supported gender specific interventions to improve health, mental health and/or legal outcomes among juvenile justice girls are lacking. The objective of this Stage II treatment trial is therefore to test the efficacy of a pre-existing, widely disseminated gender-responsive drug use treatment (VOICES) among 130 girls who are at-risk for or already involved with the justice system. We seek to test the effect of VOICES on girls' drug and alcohol use, HIV/STI risk, psychiatric symptoms and recidivism as well as explore moderators and mediators of outcomes. Girls and young women, ages 12-24 (N= 6 juveniles for Phase I Intervention Run-Through; N=130 for Phase II RCT study) will be recruited from justice partners (probation, diversion programs) and school partners (high schools/middle schools). Participants will be randomized to either the VOICES (active) intervention (n=65) or a Girl Health (attention control) condition (n=65). In Phase I (first six months of Year 1), 6 juveniles will be recruited to complete the Intervention Run-Through and research assessment once to allow testing of RCT intervention and assessment procedures prior to the RCT phase. In Phase II (last half of Year 1 through Year 4), 130 girls will be recruited and randomized at baseline and then re-assessed at mid-treatment, end of treatment, 3 months and 6 months post-intervention. Biological specimens for juvenile drug use will also be collected at each 3-month assessment. Efficacy trial results can be used to make immediate changes to current widespread program delivery resulting in direct impact on the field of evidence-based gender-responsive substance use interventions for juvenile justice girls and young women.

ELIGIBILITY:
Inclusion Criteria:

130 court-involved, non-incarcerated (CINI) female juvenile offenders or those at-risk for court-involvement, ages 12-24, who report any alcohol, marijuana or other drug use in the past 90 days will be eligible for enrollment with the following criteria:

1) Determined to be in need of substance use treatment by the court intake worker, probation officer, presiding judge or magistrate, and/or school counselor; 2) Legal guardian available to consent for child's participation, if the child is under the age of 18, and 3) Child is English speaking.

Exclusion Criteria:

1. meet DSM-V criteria for substance use disorder with current severity rating of severe (6 or more symptoms) (as determined through referral partner);
2. already in substance use treatment (residential or outpatient) and wish to remain with outside provider (as determined through referral partner);
3. observable cognitive or developmental delays or active psychosis that would interfere with completing consent, assessment or intervention.

Ages: 12 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — To be eligible for the study, participants must be female-identified
Enrollment: 132 (Actual)
Dates: Start 2014-09; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Marijuana Use | baseline, 1-month post-baseline (mid-treatment), 3 months post-baseline (end of treatment), and -3 and -6 month post-treatment completion to assess change over time
  self-reported frequency (e.g., number of days used) as measured by the Adolescent Risk Behavior Assessment (ARBA)
Alcohol Use | baseline, 1-month post-baseline (mid-treatment), 3 months post-baseline (end of treatment), and -3 and -6 month post-treatment completion to assess change over time
  self-reported quantity and frequency (e.g., number of days used, number of drinks consumed each day) as measured by the Adolescent Risk Behavior Assessment (ARBA)
Other Drug Use | baseline, 1-month post-baseline (mid-treatment), 3 months post-baseline (end of treatment), and -3 and -6 month post-treatment completion to assess change over time
  self-reported quantity and frequency (e.g., number of days and types of other drugs used) as measured by the Adolescent Risk Behavior Assessment (ARBA)
Drug Urinalysis Screen | baseline, 3 months post-baseline (end of treatment), and -3 and -6 month post-treatment completion to assess change over time
  Collateral measure of recent substance use (10-panel screen for Methadone, Amphetamine, Opiate, Oxycodone, Benzodiazepines, Barbiturates, Methamphetamine, Cocaine, Marijuana and Propoxyphene)
HIV/STI risk behavior | baseline, 1-month post-baseline (mid-treatment), 3 months post-baseline (end of treatment), and -3 and -6 month post-treatment completion to assess change over time
  self-reported frequency of sexual activity, condom use at last sex and substance use during sexual activity measured by the Adolescent Risk Behavior Assessment (ARBA)

SECONDARY OUTCOMES:
Psychiatric Symptoms | baseline, 1-month post-baseline (mid-treatment), 3 months post-baseline (end of treatment), and -3 and -6 month post-treatment completion to assess change over time
  Brief Symptom Inventory (self-report psychiatric symptom questionnaire)
Traumatic Stress | baseline, 1-month post-baseline (mid-treatment), 3 months post-baseline (end of treatment), and -3 and -6 month post-treatment completion to assess change over time
  National Stressful Events Survey PTSD Short Scale (NSESSS; self-report of posttraumatic stress symptoms and severity)
Recidivism | baseline to 6-months post-treatment completion
  Collateral/legal chart data to measure whether youth accrues any new/additional legal charges, is arrested and/or detained

CONTACTS AND LOCATIONS:
Overall Officials: Marina Tolou-Shams, Ph.D., Principal Investigator — UC San Francisco
Locations (1):
- UCSF Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramos LMC, Delgadillo J, Velez S, Dauria E, Salas J, Tolou-Shams M. Collecting Social Media Information in a Substance Use Intervention Trial With Adolescent Girls With Lifetime Substance Use History: Observational Study. JMIR Form Res. 2021 Sep 10;5(9):e25405. doi: 10.2196/25405. PMID 34505833